CLINICAL TRIAL: NCT07312435
Title: B-vitamins and ω-3 Fatty Acids to Modulate Brain Ageing in European Citizens Through Improved Nutrition: the BOOMERANG Project
Brief Title: B-vitamins and Omega-3 Fatty Acids and Biomarkers of Brain Atrophy.
Acronym: BOOMERANG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Maastricht University (Other); University of Dublin, Trinity College (Other); Aker BioMarine (Unknown); University of Ulster (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Stine Marie Ulven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REK sør-øst A 912838
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Cognitive Function
Keywords: Nutrition; Omega3; B vitamins; older adults; cognition
MeSH Terms: conditions — Dementia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive daily supplementation of one pill of B-vitamins (0.5 mg B12, 0.8 mg folate, 10 mg B6 and 10 mg riboflavin) + six pills of 500 mg Lysoveta, in total 3 g Lysoveta (480 mg EPA, 240 mg DHA).
  Interventions: Dietary Supplement: Intervention
- Control (Placebo Comparator): The control group will receive daily supplementation of one placebo pill matching the B-vitamins and one placebo pill matching Lysoveta.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Intervention — The intervention group will receive daily supplementation of one pill of B-vitamins (0.5 mg B12, 0.8 mg folate, 10 mg B6 and 10 mg riboflavin) + six pills of 500 mg Lysoveta, in total 3 g Lysoveta (480 mg EPA, 240 mg DHA). Lysoveta is an LPC-bound EPA/DHA supplement from krill which Aker BioMarine has recently developed.
  Arms: Intervention
Other: Control — The control group will receive daily supplementation of one placebo pill matching the B-vitamins and one placebo pill matching Lysoveta. the placebo capsules will contain 500 mg of mixed vegetable oil (comprising a blend of olive-, maize-, and palm kernel oil and medium-chain triglycerides, in a ratio of 4:4:3:2)
  Arms: Control

SUMMARY:
A poor nutrition status is a modifiable risk factor for cognitive decline and dementia. In particular, evidence links low status of certain B-vitamins and ω-3 fatty acids (ω-3 FA) with a greater risk of cognitive decline and dementia. Although these dietary components are typically investigated separately, post-hoc analyses of existing clinical trial data and experimental work indicate that B-vitamins and ω-3 FA may exert synergistic beneficial effects on processes related to brain health and cognition. However, this combination has not been tested directly in humans. In the proposed BOOMERANG project, we will study the effects of jointly supplementing with B-vitamins and a highly bioavailable ω-3 FA supplement, Lysoveta, on a robust biomarker of brain atrophy, the neurofilament light chain, in a double-blinded randomized controlled trial (RCT) over 3 months in older adults. We will also examine the secondary effects of the supplement of quality of life and cognitive function.

DETAILED DESCRIPTION:
We will assess the effects of combined supplementation of B-vitamins and omega-3 fatty acids on neurofilament light chain (NfL), a biomarker of brain atrophy, in a group of older adults. The primary outcome is the change in plasma NfL, which is a marker related to inflammation, brain atrophy, and worsening of cognitive performance. The secondary outcomes are related to change in plasma homocysteine, B-vitamins, EPA, DHA, omega-3 index (the percentage of EPA and DHA in red blood cells), and biological age using epigenetic markers. These are biomarkers that can tell us about the effect of the supplement in the body. We also want to study the effect of the intervention on gene expression profiles and metabolite profiles. In addition, we will include secondary outcome measures of quality of life (SF-36) that include affective symptoms, as these can be a forerunner to developing cognitive impairment. We are also collecting data on their cognitive performance, as this is related to brain atrophy and neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* A low baseline B-vitamin status as assessed by plasma tHcy > 11 μmol/L
* Normal MMSE score (>25)

Exclusion Criteria:

* Unable to give informed consent
* Fatty fish intake > 2 times per week
* daily omega-3 supplementation
* daily B-vitamin supplementation
* history of B12-injections
* Serum creatinine > 90 μmol/L for women and > 105 μmol/L for men (above reference values)
* aspirin use
* renal disease
* active cancer
* Participants can be included if they accept to not take omega-3 supplementation or B-vitamin supplements during the study. They should stop using it and wait 12 weeks before they are invited to a screening visit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Neurofilament light chain (NfL) | 3 months
  To assess the effects of combined supplementation of B-vitamins and omega-3 fatty acids on neurofilament light chain (NfL), a biomarker of brain atrophy in a group of elderly

SECONDARY OUTCOMES:
Cognitive function | 3 months
  Neuropsychological tests of global and domain specific cognitive functions will be assessed using a test battery that includes the Mini-Mental state Examination, Cognistat, and Cerad test battery (working memory, verbal fluency, constructional praxis).
Change in plasma homocysteine | 3 months
  Change in plasma homocysteine
B-vitamins | 3 months
  B-vitamins (B12, folate, B6 and riboflavin)
Omega-3 | 3 months
  EPA, DHA, omega-3 index (the percentage of EPA and DHA in red blood cells)

OTHER OUTCOMES:
Biological age | 3 months
  Biological age using epigenetic clocks
Biomarkers of brain atrophy, | 3 months
  p-tau, inflammation,
Quality of life in older adults | 3 months
  Quality of life RAND SF-36
Transcriptome PBMC | 3 months
  Biomarker
Metabolome in plasma | 3 months
  Biomarker
Gut microbiome | 3 months
  Biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Institute of Basic Medical Sciences, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
We are not allowed to share IP data due to the Univerity of Oslos data protection and regional ethical comittee rules.